CLINICAL TRIAL: NCT00541398
Title: Antipsychotic Polypharmacy: Prevalence, Background and Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: National Board of Health, Denmark (Other Government)
Responsible Party: Professor Birte Glenthøj, Center for Neuropsychiatric Schizophrenia Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0-204-03-9-9
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
Keywords: Antipsychotic polypharmacy; Schizophrenia; Implementation of clinical guidelines
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Behavioral: Implementation of guideline
- B (No Intervention)

INTERVENTIONS:
Behavioral: Implementation of guideline — Outreach visits with interactive education for health staff
  Arms: A

SUMMARY:
The primary purpose of the study is to investigate whether an intensive educational intervention can reduce the use of antipsychotic polypharmacy. It is hypothesised that the use of antipsychotic polypharmacy is, in some degree, dependent on non-patient related factors.

DETAILED DESCRIPTION:
Several surveys have shown a high prevalence of antipsychotic polypharmacy (concomitant prescription of at least 2 different antipsychotics) among patients with schizophrenia even though international guidelines recommend monotherapy.

From register data areas with differences in the prevalence of antipsychotic polypharmacy will be identified. Two high prevalence areas will be randomized to either control or intervention area. In the intervention area an intensive educational intervention consisting of outreach visits with a multifaceted approach will be carried out with the duration of 1 year.

Differences in health staff related factors such as knowledge and attitude towards clinical guidelines will be assessed with a questionnaire before and after the intervention in the intervention area as well as in the low prevalence area at baseline.

Medical records data describing the use of antipsychotic polypharmacy will be collected. With register data health economic issues will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The intervention is not aimed directly to the patients but their health care providers.
* Patients with schizophrenia (F2* diagnosis according to ICD-10) taking antipsychotic medication and their health care providers in the specified areas will enter the study:
* The patients will enter with data from their medical record, register data and a few exploring interviews while the health staff will enter with their questionnaire data.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of antipsychotic polypharmacy | 1 year

SECONDARY OUTCOMES:
Questionnaire assessment of non-patient related factors. Medical records data. Cost-effectiveness analysis. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthøj, Professor, Study Director — University of Copenhagen
Locations (1):
- CNSR, Glostrup Municipality, Denmark